CLINICAL TRIAL: NCT06345924
Title: Meraki: Music Therapy Protocol for People with Palliative Care
Brief Title: Music Therapy for Cancer Patients(Meraki_PC)
Acronym: Meraki_Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, M. Antonia Pérez-Marín, Associate Professor, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Meraki_Palliative Care
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Palliative Care
Keywords: cancer; psychological intervention; palliative care; music therapy-based treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Patients who receive the treatment program, will previously constitute their own control group (waiting list control group).
- Experimental group (Experimental): The study will commence with an initial evaluation (T1) one week after the patients' admission to the hospital. After an equal amount of time has passed without receiving any treatment, patients will undergo a re-evaluation (T2). Subsequently, patients will receive the music therapy treatment protocol, which consists of three sessions. Finally, patients will undergo a third evaluation (T3) after completing the treatment. Patients will undergo assessment before and after each music therapy session. Before the session, they will report their physical and emotional state, as well as their memory of the previous session's effects. After the session, they will be evaluated on their physical and emotional state, as well as the perceived effects of the current session. The therapy will consist of three individual sessions.
  Interventions: Behavioral: MERAKI_PC

INTERVENTIONS:
Behavioral: MERAKI_PC — The three music therapy sessions focus on helping the patient to adjust to their situation. The aim is to provide emotional support and encourage communication between family members through music. In addition, the therapy will help the patient to appreciate their remaining abilities and encourage their involvement in the rehabilitation process. The second session focuses on living in the present through re-identification. The session aims to improve the symptoms associated with the illness by focusing on the present situation and encouraging expression.
  The main aim of the final session, 'The Journey of Life - Leaving a Mark', is to recapitulate and provide support.
  Songs are used during the session, taking into account musical preferences.
  Arms: Experimental group

SUMMARY:
The overall aim of the study is to analyse the impact of a music therapy-based treatment on the emotional well-being and quality of life of cancer patients in palliative care (PC). To this end, the effectiveness and efficiency of a music therapy-based treatment to improve adaptation to illness and psychological well-being in this population will be validated and implemented.

Specifically, the implementation of an individualised treatment programme for palliative care patients will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* The patient is receiving palliative care for an oncological diagnosis and was admitted to the hospital a week ago. They do not have moderate to severe cognitive impairment. This treatment is for oncological patients in an advanced stage who are receiving palliative anti-tumour treatment such as chemotherapy and/or radiotherapy. These patients require support treatment that cannot be provided at home due to their complexity. The patient is in an advanced or terminal phase of the disease according to WHO criteria.
* Be over 18 years of age.
* Have preserved cognitive ability (SPMSQ, Pfeiffer). More than 2 errors (3 in illiterate persons) would suggest the presence of cognitive impairment.
* Have signed the informed consent form
* Have completed at least 2 of the 3 treatment sessions and have completed the pre-test and post-test assessment.

Exclusion Criteria:

-Estimated survival time. Patients with a life expectancy of two weeks or less shall not be operated on.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety and Depression Symptomatology (T1, T2 and T4) | Baseline up to 1 month
  HADS: This instrument evaluates affective disorders in non-psychiatric hospital settings. It comprises 14 items with a 4-point Likert-type response format (ranging from 0 to 3). Higher scores indicate more severe symptoms of anxiety and depression.
Change in Quality of Life (T1, T2 and T4) | Baseline up to 1 month
  EORTC QLQ-C30. It is the most widely used quality of life questionnaire in clinical trials in Europe. It is a cancer-specific questionnaire consisting of 30 items assessing quality of life. Higher scores indicate poorer quality of life for patients.
Change in emotional distress (T1, T2, T3 and T4) | Baseline up to 1 month
  The patient's overall rating of emotional distress (distress) experienced can be measured using a single-item visual analogue scale that scores from 0 to 10.

SECONDARY OUTCOMES:
Change in Social Suport (T1 and T4) | Baseline up to 1 month
  MOS: is the most appropriate instrument available in daily practice to study and evaluate social suport. By means of 20 items, it provides information on the emotional, instrumental, affective and positive social interaction dimensions, as well as offering an overall index of social support. A higher score indicates more social support.
Change in Resilience (T1 and T4) | Baseline up to 1 month
  Brief Resilient Coping Scale. This is a 4-item scale adapted to the Spanish context. Each item is scored on a 5-point scale, from 1 ("strongly agree") to 5 ("strongly disagree"). Higher scores reflect greater resilience.
Change in Spirituality (T1 and T4) | Baseline up to 1 month
  GES questionnaire: this instrument is composed of 6 open-ended questions designed to facilitate trust and disclosure of the patient, his biography and inner world, followed by 8 items assessing spirituality as a general factor through 3 spiritual dimensions: intrapersonal, interpersonal and transpersonal. The patient responds by indicating the extent to which they identify with the items, with answers ranging from 0 (indicating 'not at all') to 4 (indicating 'very much'). A higher score indicates a greater feeling of spirituality.
Change Knowledge of the disease (T1 and T4) | Baseline up to 1 month
  Clinician's assessment of the degree of acceptance, understanding, response difficulties and perception of the potential benefits of the application of the tool to patients.
Barthel Index | Baseline
  The purpose of this assessment is to evaluate the patient's functional independence. It involves assessing their ability to perform 10 activities of daily living, including eating, washing, dressing, grooming, bowel movements, urination, toileting, transferring, ambulation, and stair use. The scores range from 0, indicating maximum dependence, to 100, indicating maximum independence.
Pfeiffer Short Form Mental State Questionnaire, SPMSQ | Baseline
  This assessment evaluates cognitive impairment through a series of 10 questions that explore orientation, remote and working memory, as well as calculation skills. Each incorrectly answered question adds one point, and more than 2 errors suggest the presence of cognitive impairment that requires further study.
Charlson Comorbidity Index (CCI) | Baseline
  This tool predicts the one-year mortality rate for patients with various comorbid conditions, including heart disease, AIDS, and cancer (a total of 8 conditions in the short version). The measure assigns a score to each condition based on the associated risk of death. A score of 0 to 1 indicates no comorbidity, 2 points indicates low comorbidity, and 3 points or more indicates high comorbidity. The total score predicts mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Marián Pérez Marín, PhD, Principal Investigator — University of Valencia
Locations (1):
- Hospital Dr. Moliner, Serra, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No